CLINICAL TRIAL: NCT00896610
Title: Natural History of Autoimmune Diabetes and Its Complications
Status: Terminated | Type: Observational
Why Stopped: All analysis with identifiable specimens/data is complete or site has no identifiers linked to the specimens/data
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090140; 09-DK-0140
Record Dates: First submitted 2009-05-08; First posted 2009-05-11 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus Type 1; Diabetes Mellitus Type 2
Keywords: Diabetes Type II; Diabetes Type 1; Autoimmunity; Type 1 Diabetes; Type 2 Diabetes; Autoimmune Diabetes; At Risk Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Diabetes: Individuals who have been diagnosed with or are at risk for developing diabetes

SUMMARY:
Background:

* Diabetes is a disease defined by abnormally high blood sugar (glucose) levels. Glucose is an essential source of energy for the body s cells, but insulin is required to move the glucose into the cells. Insulin is a hormone produced by the pancreas that allows glucose to enter cells.
* In diabetes, the body is unable to supply enough insulin to meet its demands. The problem may be a low supply of insulin or a high demand for insulin. Someone who has been diagnosed with diabetes has lost much of their insulin-producing capacity. Clinical studies have shown that good control of blood sugar is essential to prevent diabetes complications like damage to the eyes, kidneys, nerves, and blood vessels.

Objectives:

* To establish a relationship with several individuals with diabetes caused by the immune system attacking the body s insulin-producing cells in order to:
* Explore why the immune system attacks insulin-producing cells.
* Understand why some individuals develop diabetes-related complications and others do not.
* Develop therapies to improve how patients can control their blood sugar levels.
* Continue to follow subjects who have completed or are considering other NIH diabetes-related studies.
* To develop improved tests for determining an individual s risk for developing diabetes and/or to accurately diagnose the exact type of diabetes.

Eligibility:

* Individuals who have been diagnosed with or are at risk for developing diabetes.

Design:

* Standard physical examination and clinical tests to determine if the patient has diabetes or to confirm a particular type of diabetes:
* None of the treatment in this study is experimental.
* Patients will receive a separate consent form for any special tests needed to learn more about their particular type of diabetes.
* Patients may be asked to provide additional urine and blood samples for use in laboratory research about diabetes.
* Researchers may offer medical treatment advice for diabetes, or explain how to improve patients diabetes management skills.

DETAILED DESCRIPTION:
Individuals with known or suspected autoimmune mediated diabetes, or healthy individuals at risk for developing the disease, will be evaluated at the NIH Clinical Center. Studies will include characterizing the disease s clinical and laboratory features, observing the natural history of the disease and its complications, evaluating responses to standard treatments. Protocol enrollees may be asked to contribute blood and/or urine samples for immunological research studies, and/or for studies designed to find parameters that increase a subject s risk for diabetes and/or its associated complications.

ELIGIBILITY:
-INCLUSION CRITERIA:

i. Clinical diagnosis of diabetes, either type 1 (T1D) or insulin-requiring type 2 (T2D),

ii. Healthy individuals who may be at risk for developing diabetes,

iii. Individuals with suspected immune mediated diabetes,

iv. Willingness of the patient or guardian to give informed consent and assent.

EXCLUSION CRITERIA:

i. Concomitant medical problems which would confound the interpretation studies of the autoimmune beta cell destructive process

ii. Concomitant medical, surgical, or other conditions for which adequate facilities or funds are not available to support their care at the NIH.

iii. Any other co-existing condition/circumstances that would make a subject unsuitable to participate in the study, as deemed by the investigators.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who have been diagnosed with or are at risk for developing diabetes
Sampling Method: Non-Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2009-05-13 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Blood glucose level | every 3 months
  Blood glucose level within a range appropriate for the patient's condition.

CONTACTS AND LOCATIONS:
Overall Officials: Ranganath Muniyappa, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Harlan DM, von Herrath M. Immune intervention with anti-CD3 in diabetes. Nat Med. 2005 Jul;11(7):716-8. doi: 10.1038/nm0705-716. No abstract available. PMID 16015359
- [Background] Haines L, Wan KC, Lynn R, Barrett TG, Shield JP. Rising incidence of type 2 diabetes in children in the U.K. Diabetes Care. 2007 May;30(5):1097-101. doi: 10.2337/dc06-1813. Epub 2007 Jan 26. PMID 17259470
- [Background] Palmer JP, Hampe CS, Chiu H, Goel A, Brooks-Worrell BM. Is latent autoimmune diabetes in adults distinct from type 1 diabetes or just type 1 diabetes at an older age? Diabetes. 2005 Dec;54 Suppl 2:S62-7. doi: 10.2337/diabetes.54.suppl_2.s62. PMID 16306342
- [Derived] Lo B, Swafford AD, Shafer-Weaver KA, Jerome LF, Rakhlin L, Mathern DR, Callahan CA, Jiang P, Davison LJ, Stevens HE, Lucas CL, White J, von Borstel R, Todd JA, Lenardo MJ. Antibodies against insulin measured by electrochemiluminescence predicts insulitis severity and disease onset in non-obese diabetic mice and can distinguish human type 1 diabetes status. J Transl Med. 2011 Nov 28;9:203. doi: 10.1186/1479-5876-9-203. PMID 22123298
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2009-DK-0140.html